CLINICAL TRIAL: NCT03560063
Title: Does the Corin Optimised Positioning System Improve Clinical Outcome in Total Hip Arthroplasty? A Multi-centre, Two-arm Randomised Control Trial
Brief Title: The Hip Arthroplasty Positioning Improvement Study
Acronym: HAPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Corin (Industry); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRAS 216084
Record Dates: First submitted 2018-05-23; First posted 2018-06-18 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2018-05

CONDITIONS: Osteoarthritis, Hip; Osteoarthritis; Arthritis; Musculoskeletal Diseases or Conditions
Keywords: arthroplasty; dislocation; templating
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis; Arthritis; Musculoskeletal Diseases; Joint Dislocations

STUDY DESIGN:
Intervention Model Description: Participants will be recruited and randomised into the two parallel study arms. Interventional arm: total hip replacement with use of the Corin Optimised Positioning System to guide templating.
  Comparator arm: total hip replacement, guided by standard templating techniques
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants: participants in both arms will undergo total hip replacement while under general anaesthetic. Participants will not be aware of the templating method used during the total hip replacement due to the general anaesthetic, therefore will remain blinded. Wounds and dressings will be the same for both study arms. Participants in the two study arms will undergo the same pre- and post-operative imaging to prevent unmasking.
  Outcomes assessors examine patients from 3 months post-operatively. There is no risk they will know which arm the patient is in, as they will not have access to the study database.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Corin OPS arm (Experimental): Total hip replacement with use of Corin Optimised Positioning System to guide implant positioning
  Interventions: Procedure: Corin Optimised Positioning System
- Standard care arm (Active Comparator): Total hip replacement with standard templating to guide implant positioning
  Interventions: Procedure: Standard templating

INTERVENTIONS:
Procedure: Corin Optimised Positioning System — Total hip replacement with implant positioning guided by Corin Optimised Positioning System.
  The experimental and active comparator arms will use the same implants for total hip replacements. The Corin Trinity shell system will be used for the acetabular system. The Corin MiniHip, TriFit, MetaFix and TaperFit implants will be used for the femoral stem implant. Surgeons will select the implant most appropriate for each patient.
  Other Names: K171847
  Arms: Corin OPS arm
Procedure: Standard templating — Total hip replacement with implant positioning guided by standard templating. The experimental and active comparator arms will use the same implants for total hip replacements. The Corin Trinity shell system will be used for the acetabular system. The Corin MiniHip, TriFit, MetaFix and TaperFit implants will be used for the femoral stem implant. Surgeons will select the implant most appropriate for each patient.
  Other Names: Anteroposterior and lateral hip radiographs
  Arms: Standard care arm

SUMMARY:
The primary objective of this study is to determine whether the Corin Optimised Positioning System (Corin, U.K.) reduces the rate of hip dislocation at one-year post-operatively compared with standard templating in patients undergoing total hip replacement.

The secondary objectives of this study are to determine whether the Corin Optimised Positioning System (Corin, U.K.) improves functional outcomes, reduces length of hospital stay, and reduces leg length discrepancy compared with standard templating in patients undergoing total hip replacement.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common joint disease worldwide affecting an estimated 10% of males and 18% of females over 60 years of age. The resultant pain and loss of function can be debilitating and in developed countries represents a large socioeconomic burden, costing between 1% and 2.5% of gross domestic product, which currently stands at over £1.5 trillion. Total hip replacement (THR) is an effective treatment for end-stage hip arthritis; however, demand for the procedure is growing rapidly, fuelled by an ageing population and the obesity epidemic. In fact, rates of THR are predicted to rise 174% between 2005 and 2030. The current commissioning environment in developed countries means that investment in iterative improvements of existing THR implant designs are unlikely to yield either significant benefits to patients or be supported by health funders. The two principle issues that concern surgeons and patients are the longevity of implants and the ability of new technologies to minimise complications such as dislocation and infection. The James-Lind Priorities Setting Partnership, an internationally recognised patient-driven organisation, has recently identified these pre-operative and intra-operative factors as targets for improving outcome following hip and knee replacement.

One of the largest costs to healthcare providers following THR is dislocation. Although the dislocation rate reported in Joint Registries is between 1 and 3% we know that this significantly underestimates the true problem, as the majority of dislocation events are managed with closed reduction and do not result in revision surgery. It is estimated that dislocation is an order of magnitude more common than reported in Registry data. Literature estimates indicate a true dislocation prevalence of 3 to 15%. The cost of dislocation is significant as the problem is often recurrent, resulting in multiple hospital admissions. The resulting average cost for each patient who suffers a THR dislocation is around £30,000.

The factors that influence dislocation are poorly understood. Conventional surgical wisdom dictates that placing a cup in the Lewinneck 'safe zone' reduces both instability and wear. A recent study of 9784 primary THRs, however, demonstrated that 58% of patients who suffered a dislocation had implants judged to be in a safe position. This has led to suggestions that the idea of one generic 'safe zone' may be misleading; instead, there is a unique optimum position to place a cup in each patient undergoing THR, based on the unique and complex interaction of the spine and pelvis of the individual. Thus, in some patients, whilst the acetabular cup appears well positioned by conventional measures, pelvic tilt and spinal position mean that the cup is placed in a position of instability during some activities.

The Corin Optimised Positioning System (OPS) is a novel platform, designed to enable delivery of the prosthetic acetabular cup into an optimised position for every patient undergoing THR. It comprises two stages: pre-operative planning and intra-operative guidance. Pre-operatively, patients undergo dynamic imaging (computed tomography scanning and X-ray films). The information gained about the relative movements of a patient's spine, pelvis and hips are used to create a personalized physiological profile. This enables calculation of the optimized acetabular cup orientation for each individual. A unique physical guide (which falls under the definition of a custom-made device in the Medical Device Directive) is then created for each patient to fit precisely into the acetabular fossa, for use intra-operatively. Intra-operatively, the Corin OPS uses laser alignment to aid the surgeon in aligning the acetabular cup in the calculated optimised orientation. One laser is affixed to an immovable pelvic screw; the other is attached to the reverse of the acetabular cup. The target orientation of the cup is achieved when the two lasers are aligned.

The aim of this trial is to assess the efficacy of the use of the Corin Optimised Positioning System in reducing post-operative hip dislocation in patients undergoing total hip arthroplasty by comparing it with current standard templating in total hip arthroplasty. All total hip implants/components used in the study will be produced by Corin for uniformity and have the required approvals. There is currently no evidence that this novel approach to templating has an effect on dislocation rate. This project aims to provide evidence that this new technique can improve outcomes for patients and have the potential to reduce the need for complex, expensive revision surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial
* Diagnosed with hip OA, post-traumatic OA, inflammatory arthropathy, avascular necrosis, or congenital or developmental hip disease, avascular necrosis of the hip
* Listed for total hip arthroplasty at one of participating centres
* Participant is fit to undergo total hip arthroplasty based on consultant anaesthetist review
* In the Investigator's opinion, is able and willing to comply with all trial requirements
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial
* Female participants of child bearing potential must be willing to ensure that they use effective contraception during the trial

Exclusion Criteria:

* Inability to provide informed consent
* Previous surgery to the ipsilateral hip
* Significant co-morbidities that would make follow up difficult or uncomfortable
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Dislocation rate | 12 months
  Incidence of hip dislocation within 12 months post-operatively

SECONDARY OUTCOMES:
Change in Harris Hip Score | Measured pre-operatively (baseline) and at 3, 6 and 12 months post-operatively
  A clinician recorded outcome score to assess functional improvement.
Change in Oxford Hip Score | Measured pre-operatively (baseline) and at 3, 6 and 12 months post-operatively
  A patient reported outcome measure (PROM) to assess patient benefit
Change in Hip and Groin Outcome Score | Measured pre-operatively (baseline) and at 3, 6 and 12 months post-operatively
  A PROM to assess patient benefit
Change in International Hip Outcome Tool 33 (iHOT33) Score | Measured pre-operatively (baseline) and at 3, 6 and 12 months post-operatively
  A PROM to assess patient benefit
Change in EuroQol 5 dimension (EQ5D) Score | Measured pre-operatively (baseline) and at 3, 6 and 12 months post-operatively
  A PROM to assess patient benefit
Change in University of California, Los Angeles (UCLA) Activity Score | Measured pre-operatively (baseline) and at 3, 6 and 12 months post-operatively
  A PROM to assess patient benefit
Change in Forgotten Joint Score | Measured pre-operatively (baseline) and at 3, 6 and 12 months post-operatively
  A PROM to assess patient benefit
Length of hospital stay | Through study completion, an average of 1 year
  Measurement of the length of the hospital admission for the total hip replacement. Measured in days.
Operation duration | Through study completion, an average of 1 year
  Measurement of the length of time of the total hip replacement operation. Measured in minutes.
Discrepancy in leg length | Measured pre-operatively and at 12 months post-operatively
  Assessment for correction in discrepancy in true leg length from pre-operative to post-operative. Measured in cm

CONTACTS AND LOCATIONS:
Overall Officials: Sion Glyn-Jones, DPhil FRCS, Principal Investigator — University of Oxford
Locations (1):
- Nuffield Orthopaedic Centre, Oxford University Hospitals Trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by the trial steering committee. Requestors will be required to sign a data access agreement

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT03560063/Prot_SAP_002.pdf